CLINICAL TRIAL: NCT07179796
Title: Digital Physical Activity Programs: a Large Scale Prospective, Observational Study
Brief Title: Digital Physical Activity Program
Status: Enrolling by invitation | Type: Observational
Sponsor: Sword Health, SA (Industry)
Responsible Party: Sponsor
Other Study IDs: SH-OBS-MV-US-01
Record Dates: First submitted 2025-09-10; First posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Overall Health; Wellbeing; Quality of Life; Mental Health
MeSH Terms: conditions — Psychological Well-Being | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observation: These programs will cover all participants interested in improving their health and wellness through increased physical activity.
  Interventions: Behavioral: Observation

INTERVENTIONS:
Behavioral: Observation — Personalized physical activity program tailored to each participant, with variations in frequency, duration, and type of activity based on their preferences, goals, fitness level, and physical ability.

SUMMARY:
The purpose of this study is to create a research repository, composed of data collected during a digital physical activity program delivered by Sword Move to individuals undergoing those programs. Sword Move intends to increase physical activity levels to stimulate the adoption of healthier, more active lifestyles. This will allow investigators to observe the effects of participants' engagement in physical activity on a variety of health and wellness based outcomes.

DETAILED DESCRIPTION:
Purpose This patient registry was designed as a research repository, composed of data collected during a digital physical activity program delivered by Sword Move to individuals undergoing those programs.

This data will allow the researchers to:

1. Assess the adoption, engagement and feasibility of digital physical activity programs to increase physical activity and its subsequent effect on health and wellness;
2. Assess the results of digital physical activity programs and compare the costs with the benefits obtained;
3. Correlate the results with patient's demographic and health condition profiles; Increase the knowledge regarding physical activity and its resultant effect on mental and physical health metrics;
4. Develop new or improved tools designed to help people improve physical activity levels and adopt healthier lifestyles.

Design Prospective, observational study

Study population These programs will cover all participants interested in improving their health and wellness through increased physical activity.

Participants will be going through a personalized physical activity program tailored to each participant, with variations in frequency, duration, and type of activity based on their preferences, goals, fitness level, and physical ability.

Outcomes The primary outcome will be the participant's progress along the program. Depending on the condition, primary and secondary outcome measures vary, but the registry will include, in all cases, a complete characterization of the participant's physical health status, as well as the periodic assessment of: a) performance indicators (through condition-specific tests); b) patient-reported outcomes (obtained using internationally validated pathology-specific questionnaires); c) compliance; d) patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* healthy individuals, or individuals with pre-existing conditions who are able to perform unsupervised exercise, unless contraindicated by their treating physician;
* older than the age of majority in their state of residence (US based);
* participant is able to understand study procedures and willing to provide informed consent.

Exclusion Criteria:

* younger than the age of majority in their state of residence;
* pain scores exceeds 6/10 on an 11-point numerical rating scale or member reports irregular movement patterns;
* undergone a surgical procedure within the last three months;
* presence of exertional red flags, as defined by the American College of Sports Medicine, and the participant has not been cleared to engage in an unsupervised exercise based program by their treating physician;
* health condition incompatible with an unsupervised exercise based program that has not been cleared by their treating physician;
* active cancer diagnosis, or is receiving treatment for cancer, and not been cleared by their treating physician to engage in an unsupervised exercise program;
* history of unexplained falls or utilization of an assistive device and has not been cleared by their treating physician to engage in an unsupervised exercise program;
* currently pregnant and has not been cleared by their treating physician to engage in an unsupervised exercise program;
* cognitive condition that prevents participant from understanding and independently executing an unsupervised exercise program.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: These programs will cover all participants interested in improving their health and wellness through increased physical activity.
Sampling Method: Non-Probability Sample
Enrollment: 300000 (Estimated)
Dates: Start 2025-09-09 (Actual); Primary Completion 2035-09 (Estimated); Study Completion 2035-12 (Estimated)

PRIMARY OUTCOMES:
Member Progress (PGIC) | Assessed at regular intervals (after 5, 9, 15, and every 6 days with activity until 3 months). Additional follow-up assessments may be undertaken at other times: 3, 6, and 12 months.
  Measured through the Patient Global Impression of Change (PGIC) questionnaire. Scores reflect the participant's perceived overall improvement (range 1-7), with higher scores indicating greater improvement.

SECONDARY OUTCOMES:
Anxiety | Assessed at baseline (upon initiation of the program) and then at regular intervals (after 5, 9, 15, and every 6 days with activity until 3 months). Additional follow-up assessments may be undertaken at other times: 3, 6, and 12 months.
  Measured through the General Anxiety Disorder-7 (GAD-7), a 7-item scale (scores 0-21). Higher scores mean higher anxiety levels.
Depression | Assessed at baseline (upon initiation of the program) and then at regular intervals (after 5, 9, 15, and every 6 days with activity until 3 months). Additional follow-up assessments may be undertaken at other times: 3, 6, and 12 months.
  Measured through the Patient Health Questionnaire-9 (PHQ-9), a 9-item scale (scores 0-27). Higher scores mean higher depression levels.
Self-reported Quality of Life | Assessed at baseline (upon initiation of the program) and then at regular intervals (after 5, 9, 15, and every 6 days with activity until 3 months). Additional follow-up assessments may be undertaken at other times: 3, 6, and 12 months.
  Assessed through the question "On a scale of 0-100, how would you rate your overall health, with 0 being the worst health imaginable and 100 the best health imaginable?"
Work productivity and absenteeism | Assessed at baseline (upon initiation of the program) and then at regular intervals (after 5, 9, 15, and every 6 days with activity until 3 months). Additional follow-up assessments may be undertaken at other times: 3, 6, and 12 months.
  Measured through Work Productivity and Activity Impairment Questionnaire (WPAI) assessed by the sub-scores: WPAI overall (combining presenteeism and absenteeism), WPAI work (presenteeism), WPAI time (absenteeism) and WPAI activities (activities of daily living impairment) (scores 0-100%). Higher scores mean greater impairment.
Self-reported Fitness Level | Assessed at baseline (upon initiation of the program) and then at regular intervals (after 5, 9, 15, and every 6 days with activity until 3 months). Additional follow-up assessments may be undertaken at other times: 3, 6, and 12 months.
  Current fitness level measured through the question "How do you currently feel when performing physical activity?". Responses are rated on a 6-point ordinal scale:
  1. Very Poor: I feel physically weak and struggle with basic physical activity;
  2. Poor: I often feel tired and find physical activity challenging;
  3. Fair: I feel average and can perform basic physical activity without much difficulty;
  4. Good: I feel above average and can perform most physical activity with ease;
  5. Very Good: I feel strong and energetic when performing challenging physical activity; 6 = Excellent: I feel extremely fit, performing strenuous physical activity with ease.
Activity Level (IPAQ) | Assessed at baseline (upon initiation of the program) and then at regular intervals (after 5, 9, 15, and every 6 days with activity until 3 months). Additional follow-up assessments may be undertaken at other times: 3, 6, and 12 months.
  Measured through the International Physical Activity Questionnaire (IPAQ). The IPAQ records frequency and duration of walking, moderate-intensity activity, vigorous-intensity activity, and sedentary behavior over the previous 7 days. Responses are converted into metabolic equivalent (MET)-minutes per week and categorized as low, moderate, or high physical activity. Higher MET-minutes indicate greater levels of physical activity.
Escalation of Care | Assessed at baseline (upon initiation of the program) and then at regular intervals (after 5, 9, 15, and every 6 days with activity until 3 months). Additional follow-up assessments may be undertaken at other times: 3, 6, and 12 months.
  Assessed through the question "Given the current status of your physical health, what is your likelihood of seeking out additional care/help to support your health or wellbeing?". Responses range from "Very unlikely" to "Very likely."
Self-reported Weight | Assessed at baseline (upon initiation of the program) and then at regular intervals (after 5, 9, 15, and every 6 days with activity until 3 months). Additional follow-up assessments may be undertaken at other times: 3, 6, and 12 months.
  Self-reported body weight, recorded in pounds, at the time of assessment.
Self-reported GLP-1 Usage | Assessed at baseline (upon initiation of the program) and then at regular intervals (after 5, 9, 15, and every 6 days with activity until 3 months). Additional follow-up assessments may be undertaken at other times: 3, 6, and 12 months.
  Assessed through the question "What is your experience with GLP-1 medications (e.g., Ozempic, Mounjaro)?"
Pain (NPRS) | Assessed at baseline (upon initiation of the program) and then at regular intervals (after 5, 9, 15, and every 6 days with activity until 3 months). Additional follow-up assessments may be undertaken at other times: 3, 6, and 12 months.
  Measured by the Numerical Pain Rating Scale (NPRS) through the question "Please rate your average pain over the last 7 days" from 0 (no pain at all) to 10 (worst pain imaginable)".
Heart Rate (wearable-measured) | Assessed continuously during physical activity sessions. Summarized at regular intervals (after 5, 9, 15, and every 6 days with activity until 3 months). Additional follow-up assessments may be undertaken at other times: 3, 6, and 12 months.
  Heart rate will be measured using a wearable device during engagement in physical activity. Measurements are recorded in beats per minute (bpm).
Daily Step Count (wearable-measured) | Steps recorded daily. Outcomes summarized at regular intervals (after 5, 9, 15, and every 6 days with activity until 3 months). Additional follow-up assessments may be undertaken at other times: 3, 6, and 12 months.
  Steps will be recorded using a wearable device as the total number of steps taken within each 24-hour period. Both total and average daily step counts will be calculated.
Sleep Duration (wearable-measured) | Recorded daily. Outcomes summarized at regular intervals (after 5, 9, 15, and every 6 days with activity until 3 months). Additional follow-up assessments may be undertaken at other times: 3, 6, and 12 months.
  Sleep will be assessed using a wearable device, including the total number of minutes spent sleeping and/or in each sleep cycle. Average minutes spent sleeping and/or in each sleep cycle will also be calculated.
Daily Active Minutes (wearable-measured) | Recorded daily. Outcomes summarized at regular intervals (after 5, 9, 15, and every 6 days with activity until 3 months). Additional follow-up assessments may be undertaken at other times: 3, 6, and 12 months.
  Physical activity time will be measured using a wearable device as the total minutes of activity per 24-hour period.
Behavior Change | Assessed at regular intervals (after 5, 9, 15, and every 6 days with activity until 3 months). Additional follow-up assessments may be undertaken at other times: 3, 6, and 12 months.
  Assessed through the question "How has your level of physical activity improved since starting the Move program?" Responses are rated on a 3-point ordinal scale: 1= Lower Activity: I'm still building my routine; 2= Moderate Activity: I'm noticing improvements and staying active a few days per week; 3= Higher Activity: I feel much more active and energized, participating in physical activities most days of the week.
Physical Health Specialist Rating | Assessed at regular intervals (after 5, 9, 15, and every 6 days with activity until 3 months). Additional follow-up assessments may be undertaken at other times: 3, 6, and 12 months.
  Assessed through the question "How would you value your overall experience with your Physical Health Specialist?", with scores ranging from 1 to 5. Higher scores indicate greater experience.
Move Plan Rating | Assessed at regular intervals (after 5, 9, 15, and every 6 days with activity until 3 months). Additional follow-up assessments may be undertaken at other times: 3, 6, and 12 months.
  Assessed through the question "How would you value your Move plan so far?", with scores ranging from 1 to 5. Higher scores indicate greater value.

OTHER OUTCOMES:
Sessions performed | Through study completion, an average of 3 months
  Number of total exercise sessions performed
Total Physical Activity Time | Through study completion, an average of 3 months
  Number of minutes spent on exercise sessions (aggregated).
Average Physical Activity Time per Week | Through study completion, an average of 3 months
  Average number of minutes spent on exercise per week
Self-reported satisfaction | Assessed at regular intervals (after 5, 9, 15, and every 6 days with activity until 3 months). Additional follow-up assessments may be undertaken at other times: 3, 6, and 12 months.
  Measured through the Net Promoter Score question collected at end of program: "On a scale from 0 to 10, how likely are you to recommend SWORD's programs to a friend or family member?")

CONTACTS AND LOCATIONS:
Overall Officials: Fernando D Correia, MD, PhD, Principal Investigator — SWORD HEALTH INC
Locations (1):
- Sword Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No